CLINICAL TRIAL: NCT04447586
Title: Soft Drink Straw as an Alternative Device of Creating Positive Expiratory Pressure (PEP) in Thoracic Surgery Patients
Acronym: PEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Collaborators: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Anna Grigoriadou, Physiotherapist, University of Thessaly
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 101ΣΕ2/16-01-2020; 725/25/11/2019 (Other: Attikon Hospital)
Record Dates: First submitted 2020-06-14; First posted 2020-06-25 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Thoracic Surgery
Keywords: Soft drink straw; Alternative PEP device; Patients undergone thoracic surgery; Cough
MeSH Terms: conditions — Cough

STUDY DESIGN:
Intervention Model Description: The first part of the study was carried out by using a device consisted of a drinking straw of an inner diameter of 5mm, a disposable mouthpiece and a manometer.The sample of this part included all the volunteers.The effectiveness of each command (A:"please blow continuously so that you feel low resistance during exhalation" and B:"please blow continuously so that you feel moderate resistance during exhalation") was estimated by comparing the average of the developing pressures during exhalation attempts arose by the corresponding command with the therapeutic range of pressure.Every volunteer performed 3 attempts for each command.The outputs of the 3rd attempt were used to the study.For the second part of the study, a number of n=8 volunteers (intervention group) was selected from the total sample and was requested to exhale as indicated by the "right" command, for 3 sets of 10 repetitions, included short breaks between sets.The remaining volunteers (n=5) consisted the control group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients following Command A and B (Active Comparator): This group of patients followed the Commands A and B with this specific order, and performed 3 exhalation attempts for each command.
  Interventions: Other: Pressure measurement during exhalation through a device consisted of a drinking straw of an inner diameter of 5mm, a disposable mouthpiece and a manometer
- Patients following Command B and A (Active Comparator): This group of patients followed the Commands B and A with this specific order, and performed 3 exhalation attempts for each command.
  Interventions: Other: Pressure measurement during exhalation through a device consisted of a drinking straw of an inner diameter of 5mm, a disposable mouthpiece and a manometer
- intervention group (Active Comparator): Intervention group was requested to exhale as indicated by the "right" command, performing 3 sets of 10 repetitions.
  Interventions: Other: Pressure measurement during exhalation through an alternative PEP device/soft drink straw.
- control group (No Intervention): Did not perform exhalation attempts by the "right" command.

INTERVENTIONS:
Other: Pressure measurement during exhalation through a device consisted of a drinking straw of an inner diameter of 5mm, a disposable mouthpiece and a manometer — Participants performed exhalation attempts through a device consisted of a drinking straw of an inner diameter of 5mm, a disposable mouthpiece and a manometer, following the instructions of Command A and B (A:"please blow continuously so that you feel low resistance during exhalation" and B:"please blow continuously so that you feel moderate resistance during exhalation") in a specific order for each group. Every volunteer performed 3 attempts for each command.The outputs of the 3rd attempt were used to the study.
  Arms: Patients following Command A and B; Patients following Command B and A
Other: Pressure measurement during exhalation through an alternative PEP device/soft drink straw. — Participants were requested to exhale as indicated by the "right" command (Command A or B), for 3 sets of 10 repetitions. This procedure included short breaks between sets.
  Arms: intervention group

SUMMARY:
Is there any possibility that patients who undergone thoracic surgery could use a simple soft drink straw as an alternative PEP device? The present study was performed to test the suitability and effect of a soft drink straw as an alternative Positive Expiratory Pressure device in patients undergone thoracic surgery and includes two sub-exploratory areas.

Before and after the measurements, the volunteers' saturation, heart rate, respiratory rate, systolic and diastolic blood pressure, dyspnea, thoracotomy pain and Cough Peak Expiratory Flow was measured.

The first part of the research, that refers to the most appropriate command for exhalation from a straw of a certain inner diameter (5mm), was carried out by using a device consisted of drinking straw, disposable mouthpiece and manometer, which valued the developed pressures during the exhalation attempts. Patients did not have visual contact with the manometer. The effectiveness of two commands (Command A: "blow continuously so that you feel little resistance during exhalation" and Command B: "blow continuously so that you feel moderate resistance during exhalation") was estimated by comparing the average of the developing pressures for every command, that occur during exhalation, with the therapeutic range of pressure. This part of the study was a cross-sectional transition and every volunteer performed 3 attempts, for each command.

The second part of the research was conducted for the evaluation of the benefits of the use of a drinking straw as an alternative device. A number of n = 8 volunteers (intervention group), who were selected from the overall sample using the closed envelope method. Taking into account the results of the first part of the research, the respondents were asked to exhale as indicated by the command that was selected before, performing 3 sets of 10 repetitions, that included short breaks between sets. The remaining volunteers (n = 5) consisted the control group.

Finally, all patients were re-examined in order to measure the Cough Peak Expiratory Flow , dyspnea, pain, saturation, heart and respiratory rate, and systolic and diastolic blood pressure, after the intervention.

DETAILED DESCRIPTION:
INTRODUCTION

The use of positive expiratory pressure devices is considered beneficial in patients who have undergone abdominal and thoracic surgery with an impact on blood gas measurement values, the hospitalization length, the use of antibiotics and the pathology of the chest. Of course, there are researchers who doubt the effectiveness of the method, mainly due to the fact that it does not possibly reduce the risk of atelectasis, especially in patients who undergone cardiac surgery. However, the method is very popular in physiotherapy, and the use of alternative devices that create positive expiratory pressure, such as water bottles or gloves, is suggested, especially in cases when the access to the classic devices is not easy, mainly during the periods of crisis.

Coughing is a process that ensures the cleaning and protection of the airways. The outcome of the thoracic surgery may often depend on the quality of the patient's cough postoperatively which may put the patient at risk that could last for up to eight weeks. The effectiveness of the cough can be assessed by measuring the peak cough flow using a peak flow meter, method that many researchers in Europe and America prefer. Cough with a maximum expiratory flow over 160 L/min could ensure a safe extubation or decannulation of severely ill and postoperative patients. Therefore, if there was a way leading to cough enhancement, this could be a lifeline to the recovery of these type of patients.

PURPOSE

The present study was performed to test the suitability and effect of a soft drink straw as an alternative positive expiratory pressure device in patients undergone thoracic surgery and includes two sub-exploratory areas.

In the first one, it was investigated the most appropriate command of exhalation into a specific internal diameter straw, whereas on the other hand, it was examined the improvement of patient's overview by using the particular alternative device.

RESEARCH HYPOTHESIS

Is there any possibility of a simple soft drink straw being an alternative PEP device which could improve the cough flow of patients who undergone thoracic surgery?

METHODOLOGY

The research was approved by "ATTIKON" University General Hospital (with reference number 725/25/11/2019) and by the University of Thessaly (with reference number 101SE2/16-01-2020).

The study was performed at the Cardiac Surgery Clinic of "ATTIKON" University General Hospital and participated all the adult thoracic surgical patients, with no limit of age, from 12-02-2020 to 08-03-2020 Patients beforehand, are informed with the purpose of the study and necessarily sign the Patient Consensus Form for their participation in the study.

Sample:

The sample of present study included all adult patients that undergone thoracic surgery, with no limit of age, with a mesosternal or lateral incision, who considered hemodynamically stable, were supplied with an O2 mixture of below 50%, full-conscious, with systolic pressure below 150 cmH20. The records were carried out on the 2nd and 3rd postoperative day.

Patients with history of chronic respiratory disease, with severe symptoms, tendency to vomit, cardiac arrhythmia due to atrial fibrillation postoperatively, and patients with angina were excluded from the study. The records were carried out in the morning or at noon and were automatically stopped if patient had any difficulty, decrease in saturation ≤90, feeling of dizziness, fainting and palpitations. The number of volunteers excluded from the study was n = 4 (2 people due to dizziness during the sitting position, 1 person with a tendency to vomit before the beginning of the process and 1 person due to re-intubation before the beginning of the process).

Procedure:

All patients were beforehand informed about the purpose of the study and signed the Patient Consensus Form in order to participate the study. Data, such as age, height and weight, type of surgery and concomitant pathologies, if any, were collected. Patients' medical records were examined to verify the collected information and find any indication that could have led to their exclusion from the study. Records and measurements were begun only after consultation with patient's doctor.

Each participant was placed in a sitting position, with his popliteal region of the knees near the edge of the bed and stayed in this position for at least 2 minutes in order to be checked that he won't develop any symptom such as discoloration of the face's skin, dizziness or fainting. In case of appearance of any of the above symptoms, patient was placed back in a supine position and the procedure stopped. Patients who felt a very light dizziness detected by overview or oral evaluation, remained seated until the symptom passes and then records and measurements were started. If the symptom continued, the procedure was stopped and patient returned to the supine position.

In the first phase of the study, all volunteers' saturation and heart rate was recorded using oximeter or monitor's indications, whereas the recording of respiratory rate followed by placing one researcher's hands on the subject's epigastrium. Both systolic and diastolic blood pressure were recorded with an analog pressure gauge, as well dyspnea (calibrated using the borg scale) and thoracotomy pain, which was quantified using the numerical pain scale (Numeric Rating Scale - oral application).

The maximum expiratory flow of air during coughing was estimated with a Peak Flow Meter (PFM) device. Participants applied their lips to a disposable mouthpiece, which was connected to the PFM and followed the command "please cough hard inside the device". The value recorded through the PFM device, which was the airflow during coughing, corresponded to the Cough Peak Expiratory Flow. Patients' surgical trauma was supported by holding a pillow on the incision during cough attempts, whereas there was no visual contact with PFM.

Intervention:

The first part of the study was to investigate the most appropriate command for exhalation through a straw of a certain inner diameter (5mm) and carried out by using a device consisted of a drinking straw, a disposable mouthpiece and a manometer to quantify the developed pressures during the exhalation attempts. The sample of this part included all the volunteers. Patients did not have visual contact with the manometer. The effectiveness of each command (Command A: "please blow continuously so that you feel low resistance during exhalation" and Command B: "please blow continuously so that you feel moderate resistance during exhalation") was estimated by comparing the average of the developing pressures during exhalation attempts arose by the corresponding command with the therapeutic range of pressure (10-20 cmH2O). This part of the study was a cross-sectional transition and every volunteer performed 3 attempts for each command. The outputs of the above attempts were recorded but only the ones of the 3rd attempt were used to the study.

The second part of the study was conducted to evaluate the benefits arising from the use of a drinking straw as an alternative PEP device. A number of n = 8 volunteers (intervention group) was selected from the total sample, using the closed envelope method. The remaining volunteers (n = 5) consisted the control group. Taking into account the results of the first part of the study, intervention group was requested to exhale as indicated by the "right" command, performing 3 sets of 10 repetitions, included short breaks between sets.

After the intervention phase, all patients were re-examined to measure the Cough Peak Expiratory Flow, dyspnea, pain, saturation, heart and respiratory rate, systolic and diastolic blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergone thoracic surgery
* no limit of age
* mesosternal or lateral incision
* hemodynamically stable
* supplied with an O2 mixture of below 50%
* full-conscious
* systolic pressure below 150 cmH20
* 2nd and 3rd postoperative day.

Exclusion Criteria:

* history of chronic respiratory disease with severe symptoms
* tendency to vomit
* cardiac arrhythmia due to atrial fibrillation postoperatively
* angina
* decrease in saturation ≤90
* dizziness
* fainting
* palpitations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2020-03-08 (Actual); Study Completion 2020-03-08 (Actual)

PRIMARY OUTCOMES:
Comparison by Commands A and B | 15 minutes
  Comparison of the outcoming pressures by Commands A and B

CONTACTS AND LOCATIONS:
Overall Officials: Kostantinos Grigoriadis, Dr, Study Director — Attikon Hospital; Garyfallia Pepera, Dr, Study Chair — University of Thessaly; Dimitrios Dougenis, Prof, Study Chair — National and Kapodistrian University of Athens
Locations (1):
- Attikon Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang XY, Wang Q, Zhang S, Tan W, Wang Z, Li J. The use of a modified, oscillating positive expiratory pressure device reduced fever and length of hospital stay in patients after thoracic and upper abdominal surgery: a randomised trial. J Physiother. 2015 Jan;61(1):16-20. doi: 10.1016/j.jphys.2014.11.013. Epub 2014 Dec 19. PMID 25534580
- [Background] Urell C, Emtner M, Hedenstrom H, Tenling A, Breidenskog M, Westerdahl E. Deep breathing exercises with positive expiratory pressure at a higher rate improve oxygenation in the early period after cardiac surgery--a randomised controlled trial. Eur J Cardiothorac Surg. 2011 Jul;40(1):162-7. doi: 10.1016/j.ejcts.2010.10.018. Epub 2010 Dec 10. PMID 21146420
- [Background] Orman J, Westerdahl E. Chest physiotherapy with positive expiratory pressure breathing after abdominal and thoracic surgery: a systematic review. Acta Anaesthesiol Scand. 2010 Mar;54(3):261-7. doi: 10.1111/j.1399-6576.2009.02143.x. Epub 2009 Oct 29. PMID 19878100
- [Background] Sehlin M, Ohberg F, Johansson G, Winso O. Physiological responses to positive expiratory pressure breathing: a comparison of the PEP bottle and the PEP mask. Respir Care. 2007 Aug;52(8):1000-5. PMID 17650355
- [Background] Dagan Y, Wiser I, Weissman O, Farber N, Hundeshagen G, Winkler E, Kazula-Halabi T, Haik J. An Improvised "Blow Glove" Device Produces Similar PEP Values to a Commercial PEP Device: An Experimental Study. Physiother Can. 2014 Summer;66(3):308-12. doi: 10.3138/ptc.2013-31. PMID 25125786
- [Background] Banner AS. Cough: physiology, evaluation, and treatment. Lung. 1986;164(2):79-92. doi: 10.1007/BF02713631. No abstract available. PMID 3084882
- [Background] Johnson D, Hurst T, Thomson D, Mycyk T, Burbridge B, To T, Mayers I. Respiratory function after cardiac surgery. J Cardiothorac Vasc Anesth. 1996 Aug;10(5):571-7. doi: 10.1016/s1053-0770(96)80130-3. PMID 8841860
- [Background] Kulnik ST, MacBean V, Birring SS, Moxham J, Rafferty GF, Kalra L. Accuracy of portable devices in measuring peak cough flow. Physiol Meas. 2015 Feb;36(2):243-57. doi: 10.1088/0967-3334/36/2/243. Epub 2015 Jan 13. PMID 25582526
- [Background] Rose L, McKim D, Leasa D, Nonoyama M, Tandon A, Kaminska M, O'Connell C, Loewen A, Connolly B, Murphy P, Hart N, Road J. Monitoring Cough Effectiveness and Use of Airway Clearance Strategies: A Canadian and UK Survey. Respir Care. 2018 Dec;63(12):1506-1513. doi: 10.4187/respcare.06321. Epub 2018 Sep 11. PMID 30206128
- [Background] Winck JC, LeBlanc C, Soto JL, Plano F. The value of cough peak flow measurements in the assessment of extubation or decannulation readiness. Rev Port Pneumol (2006). 2015 Mar-Apr;21(2):94-8. doi: 10.1016/j.rppnen.2014.12.002. Epub 2015 Feb 14. PMID 25926373
- [Background] Ahmad AM. Essentials of Physiotherapy after Thoracic Surgery: What Physiotherapists Need to Know. A Narrative Review. Korean J Thorac Cardiovasc Surg. 2018 Oct;51(5):293-307. doi: 10.5090/kjtcs.2018.51.5.293. Epub 2018 Oct 5. PMID 30402388
- [Background] Holdgate A, Asha S, Craig J, Thompson J. Comparison of a verbal numeric rating scale with the visual analogue scale for the measurement of acute pain. Emerg Med (Fremantle). 2003 Oct-Dec;15(5-6):441-6. doi: 10.1046/j.1442-2026.2003.00499.x. PMID 14992058
- [Background] Fiore JF Jr, Chiavegato LD, Denehy L, Paisani DM, Faresin SM. Do directed cough maneuvers improve cough effectiveness in the early period after open heart surgery? Effect of thoracic support and maximal inspiration on cough peak expiratory flow, cough expiratory volume, and thoracic pain. Respir Care. 2008 Aug;53(8):1027-34. PMID 18655740
- [Background] Hristara-Papadopoulou A, Tsanakas J, Diomou G, Papadopoulou O. Current devices of respiratory physiotherapy. Hippokratia. 2008;12(4):211-20. PMID 19158964
- [Background] Liverani B, Nava S, Polastri M. An integrative review on the positive expiratory pressure (PEP)-bottle therapy for patients with pulmonary diseases. Physiother Res Int. 2020 Jan;25(1):e1823. doi: 10.1002/pri.1823. Epub 2019 Nov 25. PMID 31762162
- See also: Breathing exercises with positive expiratory pressure after abdominal surgery - The current physical therapy practice in Sweden — https://www.researchgate.net/publication/278282011_Breathing_exercises_with_positive_expiratory_pressure_after_abdominal_surgery_-_The_current_physical_therapy_practice_in_Sweden
- See also: Is retained mucus a risk factor for the development of postoperative atelectasis and pneumonia? -- Implications for the physiotherapist — https://www.researchgate.net/publication/239325269_Is_retained_mucus_a_risk_factor_for_the_development_of_postoperative_atelectasis_and_pneumonia_--_Implications_for_the_physiotherapist